CLINICAL TRIAL: NCT03053492
Title: Establishing the Functional Viability and Dose-response of Duck, Duck Punch: A Stroke Rehabilitation Computer Game
Brief Title: Functional Viability Duck Duck Punch
Acronym: DDPSBIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00059924; 1R44NS097061-01A1 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Rehabilitation; Recovery of Function; Stroke
Keywords: Video Games
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Stroke survivors will either play a custom designed computer game for stroke rehabilitation called Duck Duck Punch or an off the shelf computer game with their weaker arm 3 times per week for 6 weeks. Evaluations will determine whether or not one computer game improved arm movement more than the other.
Who Masked: Outcomes Assessor
Masking Description: Blinded raters perform scoring of all assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Duck Duck Punch (Experimental): Subjects in this arm will engage in Duck Duck Punch Play, a custom designed computer game developed for stroke rehabilitation for 6 weeks.
  Interventions: Device: Duck Duck Punch Play
- Commercially Available Game (Active Comparator): Subjects in this arm will engage in a Commercially Available Game Play off-the-shelf computer game for 6 weeks.
  Interventions: Behavioral: Commercially Available Game Play

INTERVENTIONS:
Device: Duck Duck Punch Play — The behavioral intervention will include playing a hands-free video game custom designed for stroke survivors.
  Arms: Duck Duck Punch
Behavioral: Commercially Available Game Play — The behavioral intervention will include playing a hands-free video game available off-the-shelf.
  Arms: Commercially Available Game

SUMMARY:
This study has 2 parts: In one part of this study, people with stroke will either play a custom designed computer game for stroke rehabilitation called Duck Duck Punch or an off the shelf computer game with their weaker arm 3 times per week for 6 weeks. Evaluations will determine whether or not one computer game improved arm movement more than the other. In the second part of the study, people with stroke, caregivers of people with stroke and stroke rehabilitation therapists will meet in several focus groups to design a useful and informative Duck Duck Punch performance report.

DETAILED DESCRIPTION:
Stroke is a problem nationally, but especially in the southeastern USA, a region known as the "stroke belt" where stroke incidence is high and age of stroke onset is low. The vast majority, >75%, of stroke survivors experience paresis of one arm/hand that does not resolve acutely. Long-term arm movement impairment restricts independence with self-care and vocational activities, increases caregiver burden and reduces quality of life. Although rehabilitation improves outcomes, systematic financial pressures increasingly limit its duration. Unfortunately, this is happening at a time when strong evidence is emerging that traditional therapy programs do not provide adequate amounts of movement practice needed for motor recovery. Thus, there is a need for innovative technology to augment traditional stroke rehabilitation programs in a way that can provide the necessary movement practice within the constraints of current rehabilitation practice.

To meet this need, the Principal Investigators developed a prototype Kinect-based post-stroke rehabilitation game called Duck Duck Punch (DDP). While maintaining the appeal of a game, DDP has a therapeutic focus because its unique design elicits an arm motor recovery process consistent with evidence-based stroke rehabilitation principles. The player moves his/her physical arm to control an avatar arm to reach and "punch" virtual ducks. Custom features allow tailoring of game difficulty to match a player's impairment level so that the player seeks to accomplish optimally challenging movement goals. By design, the avatar does not respond to atypical arm motions, which encourages the player to trial and error a variety of motions until implicitly learning the more normal strategy. Thus, unlike most commercially available "off the shelf" games, success requires "therapist approved" healthy arm motions. Success motivates continued game play for extended practice of healthy motions. Therapists can integrate DDP into in-clinic or in-home therapies for additional quasi-supervised movement practice and receive a performance report that quantifies and monitors progress toward recovery goals. Further development of this report will enable its integration into a billable rehabilitation program.

The Investigators licensed DDP and formed a company, Recovr, which has received investment funding for initial start-up and market research. Of note, DDP has also received FDA 510(k) Clearance to "support physical rehabilitation of adults in the clinic and at home via performance of therapist-assigned reach exercises for the upper extremities." In a funded NIH/NIGMS pilot project, the investigators established the technical merit and feasibility of DDP as a tool to augment inpatient, outpatient and home-based stroke rehabilitation by increasing therapist- and patient-directed movement practice opportunities. Very promising results motivated the current project that seeks to test the functional viability of DDP and determine its commercial potential.

ELIGIBILITY:
Inclusion Criteria:

* experienced unilateral hemispheric ischemic or hemorrhagic stroke at least 3 months but no more than 7 years prior
* exhibit voluntarily shoulder flexion of the affected arm ≥30° with simultaneous elbow extension ≥20°. The investigators reason that persons at this motor ability level have residual arm activation and enough ability to engage in treatment-related reaching movements elicited by the computer games
* baseline FMA-UE score of at least 19 points but no more than 52 points (out of 60 points) based on previously published research by this study's investigators in which categories were defined based on post-stroke UE motor impairment
* passive range of motion in affected shoulder, elbow and wrist within 20 degrees of normal values
* 21-90 years of age
* a caregiver or friend who is willing to assist with the set up and operation of the computer game throughout the 6 week intervention.

Exclusion Criteria:

* lesion in brainstem or cerebellum because lesions in these locations my interfere with the visual-perceptual and cognitive skills needed for motor re-learning as is expected to occur as a result of the intervention
* presence of other neurological disease that may impair motor skills (e.g., Parkinson's Disease)
* pain in the affected arm that interferes with reaching movements
* significant cognitive impairment, defined as Montreal Cognitive Assessment score < 22
* orthopedic condition or impaired corrected vision that alters the kinematics of reaching
* unable to travel to the UE Motor Function Laboratory in Charleston, South Carolina 4 times (pre-, mid- post- and retention testing).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Woodbury, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study, de-identified data will be available to other researchers and may be obtained by emailing the PI

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duck Duck Punch | Commercially Available Game
Started | 33 | 33
Completed | 25 | 27
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duck Duck Punch | Commercially Available Game | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.45 (12.33) | 58.24 (10.91) | 60.85 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 33 | 32 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 17 | 30
  White | 20 | 13 | 33
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Upper Extremity Assessment (FMA-UE)
Description: 33 item measure of upper extremity (UE) motor control impairment. Total scores were analyzed from 0/66 (indicating a severe impairment, no motor control) to 66/66 (indicating a mild impairment, with near normal motor control)
Time Frame: Change from baseline at post 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duck Duck Punch | Commercially Available Game
Number analyzed (Participants) | 33 | 33
Units on a scale | 0.13 (0.03) | 0.12 (0.04)

2. Secondary Outcome: Wolf Motor Function Test (WMFT)
Description: The Wolf Motor Function Test contains 15 items, each of which measure upper extremity functional ability by recording the time (seconds) required to accomplish the task. High functional ability is evident in quicker performance times near 0 seconds. Low functional ability is evident in slower performance times near 120 seconds. The assessment is scored by recording the time to perform each of the 15 items (0 seconds to 120 seconds per item), then the average item performance time is calculated. A small average item performance time (near 0 seconds) indicates higher functional ability and thus a better outcome. A large average item performance time (near 120 seconds) indicates less functional ability and thus a poorer outcome.
Time Frame: Change from baseline at post 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: Time (seconds)
Arm/Group | Duck Duck Punch | Commercially Available Game
Number analyzed (Participants) | 33 | 33
Time (seconds) | 0.12 (0.10) | -0.5 (0.14)

3. Secondary Outcome: Kinematic Variable; Shoulder Flexion-elbow Extension Interjoint Coordination
Description: Shoulder flexion-elbow extension interjoint coordination. Correlation between the shoulder flexion and elbow extension joint angles during a forward reach movement. Values range from -1 (indicating an abnormal flexor synergy pattern, i.e. higher impairment) to 1 (indicating movement similar to a healthy individual, i.e. lower impairment).
Time Frame: Change from baseline at post 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Duck Duck Punch | Commercially Available Game
Number analyzed (Participants) | 33 | 33
Units on a scale | -0.02 (0.20) | -0.01 (0.18)

4. Secondary Outcome: Kinematic Variable; Trunk Displacement
Description: Displacement of the upper trunk marker during reaching task
Time Frame: Change from baseline at post 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Duck Duck Punch | Commercially Available Game
Number analyzed (Participants) | 33 | 33
mm | 13.89 (38.84) | -6.02 (23.73)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of the study a total of 1 year, and 11 months.
Arm/Group | Duck Duck Punch | Commercially Available Game
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 1/33 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duck Duck Punch (N=33) | Commercially Available Game (N=33)
Fall Unrelated to Study (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Visit to ER Unrelated to Study (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03053492/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03053492/SAP_001.pdf